CLINICAL TRIAL: NCT03157024
Title: Validation of a Newly Developed Sham Press Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Hyangsook Lee, KMD, PhD, Professor, Kyunghee University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: KHSIRB-16-009
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Press Needle - Ring Sham (RS) (Experimental): A sterilised stainless steel press needle that only has the ring-shaped head of needle without needle body has three layers of adhesive tape. Between the first and second layer is the head of needle to support needle body while maintaining identical appearance and the third layer is attached to skin. RS will be placed on 1 cm medial to acupoint LI11 and ear wrist, a non-specific control auricular acupoint used in the previous literature of the non-dominant side. An acupoint detector (personal TENS electronic acupuncture, Hammtek Korea, Seoul, Korea) will be used to locate points with lower skin impedance than those nearby.
  Interventions: Device: Ring Sham (RS)
- Real Needle (RN) (Active Comparator): A sterilised stainless steel press needle (diameter 0.18 mm X length 1.5 mm, Dongbang Acupuncture Inc., Boryeong, Chungcheongnam-do, Korea) has three layers of adhesive tape. Between the first and second layer is the head of needle to support needle body and the third layer is attached to skin. RN will be placed on acupoint LI11 and ear shenmen of the non-dominant side. An acupoint detector (personal TENS electronic acupuncture, Hammtek Korea, Seoul, Korea) will be used to locate points with lower skin impedance than those nearby.
  Interventions: Device: Real Needle (RN)
- Kim Sham (KS) (Sham Comparator): A sterilised stainless steel press needle (diameter 0.18 mm X length 1.5 mm, Dongbang Acupuncture Inc., Boryeong, Chungcheongnam-do, Korea) with a blunted tip has three layers of adhesive tape. Between the first and second layer is the head of needle to support needle body while maintaining identical appearance and the third layer is attached to skin. KS will be placed on 1 cm medial to acupoint LI11 and ear wrist, a non-specific control auricular acupoint used in the previous literature of the non-dominant side. An acupoint detector (personal TENS electronic acupuncture, Hammtek Korea, Seoul, Korea) will be used to locate points with lower skin impedance than those nearby.
  Interventions: Device: Kim Sham (KS)

INTERVENTIONS:
Device: Ring Sham (RS)
  Arms: Sham Press Needle - Ring Sham (RS)
Device: Real Needle (RN)
  Arms: Real Needle (RN)
Device: Kim Sham (KS)
  Arms: Kim Sham (KS)

SUMMARY:
This is a single blind randomised controlled trial involving healthy volunteers to determine feasibility and blinding property of two types of sham press needles.

DETAILED DESCRIPTION:
A total of 84 healthy volunteers will be recruited and randomly allocated to receive real needles (RN), previously validated Kim Sham needles (KS), or newly developed Ring Sham needles (RS) at a 1:1:1 ratio. Acupuncture sensation, blinding, and feasibility in a future clinical trial will be measured along with other physiological measurements including tactile sensitivity, interoceptive sensitivity, and electrodermal activity.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* not participating in other clinical studies at the time of study participation
* voluntary participation

Exclusion Criteria:

* not satisfying the inclusion criteria
* pregnancy or breast-feeding at the time of study participation
* open sores or skin diseases on the non-dominant elbow or ear where needles would be placed
* having taken analgesics in 24 hours before participation
* any other diseases or conditions that might prevent the participant from receiving acupuncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
Blinding property | After needling on the 1st day visit
  Blinding property will be evaluated: the participants will be asked 'which type of acupuncture do you think you have received?' and choose 1 answer out of real, sham, or don't know.

SECONDARY OUTCOMES:
Adhesive power | On the next day visit (1 day after needling)
  It will be assessed whether sham press needle remains in place for at least 2 days (yes/no).
Acupuncture sensation measured by De-qi questionnaire | After needling on the 1st day visit
  De-qi questionnaire (Kim et al.) will be used to evaluate acupuncture sensation.
Acupuncture sensation measured by De-qi questionnaire | After needle removal on the next day visit (1 day after needling)
  De-qi questionnaire (Kim et al.) will be used to evaluate acupuncture sensation.
Blinding property | After needle removal on the next day visit (1 day after needling)
  Blinding property will be evaluated: the participants will be asked 'which type of acupuncture do you think you have received?' and choose 1 answer out of real, sham, or don't know.

OTHER OUTCOMES:
Acupuncture Belief Scale (ABS) | After needling on the 1st day visit
  A Korean version of Acupuncture Belief Scale (ABS), a 36-item self-report on a 5-point Likert scale will be used to evaluate acupuncture experiences and beliefs.
Tactile sensitivity | On the 1st day visit
  Tactile sensitivity will be measured using von Frey filament.
Interoceptive sensitivity | On the 1st day visit
  Using a modified method by Schandry, the participants will be asked to count their own heartbeats with eyes closed during the three counting phases that vary in length randomly, i.e. 25, 35, and 45 seconds. Beginning and end of a phase will be given verbally by the experimenter. Information on the length of the three counting phases will not be open to participants. Heart rate will also be recorded and analysed by a computer-based data acquisition system (MP150 data acquisition system, version 4.3.0, Biopac® Systems, Inc., Goleta, CA, USA).
Electrodermal activity (EDA) | On the 1st day visit
  EDA data will be obtained to evaluate autonomic response following acupuncture needling (MP150 data acquisition system, version 4.3.0, Biopac® Systems, Inc., Goleta, CA, USA).
Acupuncture credibility | After needle removal on the next day visit (1 day after needling)
  Credibility of the acupuncture treatment will be evaluated using a credibility test by Vincent et al.

CONTACTS AND LOCATIONS:
Overall Officials: Hi-Joon Park, KMD, PhD, Study Director — Kyunghee University
Locations (1):
- Acupuncture & Meridian Science Research Centre, Kyung Hee University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim S. Creating an instrument for a successful double-blind acupuncture placebo. J Acupunct Meridian Stud. 2008 Sep;1(1):36-41. doi: 10.1016/S2005-2901(09)60005-4. Epub 2009 Mar 24. PMID 20633453
- [Background] Lee H, Bang H, Kim Y, Park J, Lee S, Lee H, Park HJ. Non-penetrating sham needle, is it an adequate sham control in acupuncture research? Complement Ther Med. 2011 Jan;19 Suppl 1:S41-8. doi: 10.1016/j.ctim.2010.12.002. Epub 2010 Dec 23. PMID 21195294
- [Background] Bang H, Ni L, Davis CE. Assessment of blinding in clinical trials. Control Clin Trials. 2004 Apr;25(2):143-56. doi: 10.1016/j.cct.2003.10.016. PMID 15020033
- [Background] Moroz A, Freed B, Tiedemann L, Bang H, Howell M, Park JJ. Blinding measured: a systematic review of randomized controlled trials of acupuncture. Evid Based Complement Alternat Med. 2013;2013:708251. doi: 10.1155/2013/708251. Epub 2013 Mar 3. PMID 23533515
- [Background] Kim Y, Park J, Lee H, Bang H, Park HJ. Content validity of an acupuncture sensation questionnaire. J Altern Complement Med. 2008 Oct;14(8):957-63. doi: 10.1089/acm.2007.0565. PMID 18925869
- [Background] Kim S, Lee S, Choi S, Park J, Kim S. Discrimination accuracy between real and sham press needles in the hands. Acupunct Med. 2015 Aug;33(4):293-8. doi: 10.1136/acupmed-2014-010678. Epub 2015 Jun 4. PMID 26044714
- [Background] Wang SM, Maranets I, Weinberg ME, Caldwell-Andrews AA, Kain ZN. Parental auricular acupuncture as an adjunct for parental presence during induction of anesthesia. Anesthesiology. 2004 Jun;100(6):1399-404. doi: 10.1097/00000542-200406000-00011. PMID 15166558
- [Background] Wang SM, Dezinno P, Lin EC, Lin H, Yue JJ, Berman MR, Braveman F, Kain ZN. Auricular acupuncture as a treatment for pregnant women who have low back and posterior pelvic pain: a pilot study. Am J Obstet Gynecol. 2009 Sep;201(3):271.e1-9. doi: 10.1016/j.ajog.2009.04.028. Epub 2009 Jun 26. PMID 19560110
- [Background] Schandry R. Heart beat perception and emotional experience. Psychophysiology. 1981 Jul;18(4):483-8. doi: 10.1111/j.1469-8986.1981.tb02486.x. No abstract available. PMID 7267933
- [Background] Vincent C, Lewith G. Placebo controls for acupuncture studies. J R Soc Med. 1995 Apr;88(4):199-202. PMID 7745565